CLINICAL TRIAL: NCT05105802
Title: Mindfulness-Based Intervention for Mild Traumatic Brain Injury
Acronym: MBI-4-mTBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Eastern Ontario (Other)
Collaborators: Mobio Interactive PTE LTD (Industry); University of Ottawa (Other); Academic Health Science Centres (Other)
Responsible Party: Principal Investigator, Andree-Anne Ledoux, Scientist, Children's Hospital of Eastern Ontario
Allocation: Not Applicable | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 20190441
Record Dates: First submitted 2021-10-08; First posted 2021-11-03 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Concussion, Mild
Keywords: mild traumatic brain injury; intervention; treatment; persistent post-concussive symptoms; quality of life; meditation
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Intervention Model Description: Double-blind randomized clinical trial with 2 groups
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double-blind study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mindfulness Intervention (Experimental): MBI training will consist of a 4-week custom-made program that include, setting intentions and check-in with mood, audio-recorded lectures, guided meditations such as body scans, and writing events journal. Each standardized course will be unlocked as the child progresses through the program. Users will be encouraged to participate in the app-based activities for a total of 10-15 minutes every day, with a minimum of 4 days in a week, over a period of 4 weeks.
  Interventions: Behavioral: Mindfulness-Based Intervention
- Cognitive Sham Application + Usual Care (Active Comparator): Usual care recommends that the patient refrain from physical and cognitive activities for 24-48 hours after injury. After the rest period, it is recommended that low to moderate levels of physical and cognitive activity be gradually started 24-48 hours after injury. The activities should be performed at a level that does not result in recurrence or exacerbation of symptoms. Children must refrain from any activities that increase the risk of re-injury (drills with body contact or that risk falls) until fully asymptomatic and cleared by their primary care or other medical provider. We consider this arm as active as participants will be assigned to a cognitive sham app (cognitive math game) delivered via the same app (same main interface as the mindfulness intervention). However, they will not take part in the MBI program for the first 4 weeks. On a daily basis, participants will be asked questions about their stress and emotions and about their symptoms.
  Interventions: Behavioral: Cognitive Sham + Usual Care

INTERVENTIONS:
Behavioral: Mindfulness-Based Intervention — Using AmDtx MBI-based app, targeted MBI training will consist of a 4-week custom-made program that include, setting intentions and check-in with mood, audio-recorded lectures, guided meditations such as body scans, and writing events journal (Appendix 5). Each standardized course will be unlocked as the child progresses through the program. Users will be encouraged to participate in the app-based activities for a total of 10-15 minutes every day, with a minimum of 4 days in a week, over a period of 4 weeks.
  Other Names: MBI, AmDtx
  Arms: Mindfulness Intervention
Behavioral: Cognitive Sham + Usual Care — Usual care recommends that the patient refrain from physical and cognitive activities for 24-48 hours after injury. After the rest period, it is recommended that low to moderate levels of physical and cognitive activity be gradually started 24-48 hours after injury. The activities should be performed at a level that does not result in recurrence or exacerbation of symptoms. Children must refrain from any activities that increase the risk of re-injury (drills with body contact or that risk falls) until fully asymptomatic and cleared by their primary care or other medical provider. The sham journey will consist of playing an open-source cognitive math game delivered through the same app as MBI, but without the mindfulness content.
  Other Names: Cognitive Sham, Usual Care
  Arms: Cognitive Sham Application + Usual Care

SUMMARY:
Mindfulness is a promising tool which may foster adaptative interpersonal qualities to reduce the risk of persistent post-concussion symptoms. The present feasibility study will customize and validate a mindfulness mobile smart-phone app easily accessible to youth and families. The study will also determine whether mindfulness training increases quality of life, reduces symptom burden and promotes neurophysiological recovery at 4 weeks post-injury in adolescents who were diagnosed with an acute concussion compared to a cognitive sham app + usual care.

DETAILED DESCRIPTION:
One in three youth with a concussion will be afflicted with persistent post-concussive symptoms (PPCS), defined as the persistence of symptoms beyond one month of injury. PPCS may impair daily activities including schoolwork, socializing, and sports, thus reducing the quality of life. Preventive psychological interventions that foster coping skills may be key to managing concussions and reducing the risk of PPCS. Mindfulness-Based Interventions (MBI) are "present-centered" interventions, encouraging acceptance of thoughts and emotions as they occur in the moment, without judgment. The goal of the present pilot and feasibility randomized clinical trial (RCT) is to investigate whether the introduction of early targeted MBI training, delivered via a mobile application, can increase the quality of life and lead to improved adaptation to acute impairments of concussion. Further, we will establish the feasibility of conducting a larger RCT by investigating the ease of recruitment, credibility score, adherence to treatment, and retention of an app-based MBI. Participants with an acute concussion will be randomly assigned to one of two groups: (1) experimental group (n=63): early introduction of the MBI training; (2) control group (n=63): sham cognitive task and usual care. The targeted MBI training consists of a 4-week custom-made program for youth. Each standardized psychoeducation of meditation practice will be unlocked as the participant progresses through the program. The curriculum is based on previous validated MBI app protocols and team expertise in MBI.

ELIGIBILITY:
Inclusion Criteria:

* Subjects presenting to CHEO's Emergency Department (ED) within 48 hours of sustaining a direct or indirect head injury
* Aged 12 through 17.99 years
* Have a concussion, as defined by the Berlin consensus statement
* Score >4 on the predicting persistent postconcussive problems in pediatric (5P) clinical rule
* Proficient in English.

Exclusion Criteria:

* Glasgow Coma Scale ≤13
* Abnormality on standard neuroimaging studies, including positive head CT findings (Note: neuroimaging is not required but may be performed if clinically indicated)
* Neurosurgical operative intervention, intubation, or intensive care required
* Multi-system injuries with treatment requiring hospital admission, operating room, or procedural sedation in ED (Note: hospital admission for observation or management of ongoing concussion symptoms is not an exclusion criteria)
* Severe chronic neurological developmental delay resulting in communication difficulties
* Intoxication at the time of ED presentation as per clinician judgment
* History of trauma as primary events (e.g., seizure, syncope, migraine)
* Prior psychiatric hospitalization
* Prior diagnosis of severe psychiatric disorder such as schizophrenia (diagnosis of anxiety or depression is not exclusionary)
* Inability to obtain a proper written informed consent/assent (e.g., language barrier, absence of parental authority, developmental delay, intoxication, patients too confused to consent)
* Legal guardian not present (certain forms need to be completed by parents/legal guardians)
* No Internet or mobile/tablet access.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 99 (Actual)
Dates: Start 2022-10-04 (Actual); Primary Completion 2024-07-06 (Actual); Study Completion 2024-07-06 (Actual)

PRIMARY OUTCOMES:
Ease of Recruitment | 48 hours post-injury
  Descriptive variable. Ease of recruitment will be defined as having at least 60% approached and eligible participants agreeing to participate. A higher score means easier recruitment.
Credibility Score (Credibility and Expectancy Questionnaire) | 1 week post-injury
  The Credibility and Expectancy Questionnaire is a 6-item The credibility score is derived from the items 1-3 and the expectancy scores is derived from the items 4-6. A higher score means better credibility. The treatment will be considered as credible if 80% of the participants rated the treatment as credible.
Retention | 4 weeks post-injury
  Descriptive variable. Adequate retention will be defined as having 70% of participants completing at least 60% of the 4-week intervention and the outcome measurement post-treatment. A higher score means better retention.
Adherence to Treatment | 4 weeks post-injury
  Calculated based on the time spent on the app. A higher score means better adherence.

SECONDARY OUTCOMES:
Pediatric Quality of Life Inventory™ version 4.0 | 4 weeks post-injury
  The Pediatric Quality of Life Inventory™ version 4.0 is a reliable and valid measure of quality of life in healthy children and adolescents and those with acute and/or chronic health conditions.The inventory covers four domains: physical, emotional, social, and school. It is a 23-item, 5-point Likert scale producing a total score (range=0-92) and 4 domain scores (physical, emotional, social, and school). Higher scores indicate better outcomes.
Health and Behaviour Inventory | 2 and 4 weeks post-injury
  The Health and Behaviour Inventory is validated symptom scale. It is a 20-item self-report questionnaire, 4-point Likert scale (total range 0-60) yielding scores for cognitive and somatic symptom scales. A higher score indicate worse outcome.
Post-Concussion Symptom Inventory (PCSI) | 2 and 4 weeks post-injury
  The Post-Concussion Symptom Inventory (PCSI) is a validated, reliable, comprehensive, self-administered instrument for children and adolescents. For the purpose of this study, the emotional and sleep domain of the PCSI adolescent scale version (20-item, 7-point Likert scale) will be used. A higher score indicate worse outcome.
Self-Efficacy Questionnaire for Children | 4 weeks post-injury
  The Self-Efficacy Questionnaire for Children is a valid and reliable assessment, Cronbach's α=0.88. It is a 24-item, 5-point Likert scale questionnaire producing a total score (0-120), and emotional, social, and academic sub-scores. A higher score indicate better outcome.
NIH Toolbox Cognitive Battery | 4 weeks post-injury
  The NIH Toolbox Cognitive Battery, a validated and reliable computerized battery designed to measure fluid cognitive functioning (executive function, attention, episodic memory, language, processing speed, and working memory). Raw performance is transformed to age-corrected standard scores, for which the normative mean in 100 and the standard deviation is 15. Other types of scores computed by the battery include fully corrected t-scores (mean of 50 and standard deviation of 10, comparing the score of the participant to those of the normative sample while adjusting for key demographic variables: age, gender, race/ethnicity, educational attainment), uncorrected standard scores (normative mean of 100 and standard deviation of 100), percentiles. Higher scores indicate better outcomes.
The Connor-Davidson Resilience Scale-10 | 4 weeks post-injury
  The Connor-Davidson Resilience Scale-10 is a validated questionnaire in an adolescent concussed population. It is a 10-item, 5-point Likert scale assessing the individual's own perception of hardiness or perceived stress (total score range=0-40). A higher score indicates better outcome.
General Anxiety Disorder 7-items (GAD) | 4 weeks post-injury
  The GAD-7 is a validated, reliable, and sensitive to treatment-related changes tool that assesses anxiety symptoms in youth. It is a 7-item, 3-point Likert scale questionnaire providing a sum score (0-21) of the level of general anxiety disorder. A higher score indicate worse outcome.
Center for Epidemiologic Studies Short Depression Scale | 4 weeks post-injury
  This is a 10-item, 4-point Likert scale questionnaire assessing the level of depression symptoms in the past week. A higher score indicate worse outcome. Total scores can range from 0 to 30. A higher score indicate worse outcome.
Child and Adolescent Mindfulness Measure | 4 weeks post-injury
  The Child and Adolescent Mindfulness Measure is a validated, 10-item, 5-point Likert scale questionnaire. A higher score indicate better outcome.
Functional Connectivity measured by Resting-State Functional MRI | 72 hours and 4th week post-injury
  A subset of 60 participants will undergo a magnetic resonance imaging scan (MRI), which includes a resting-state functional MRI to assess function connectivity. To measure intra- and interconnectivity between regions of interest (default-mode network) and regions across the brain, will be measured. To calculate functional connectivity per participant, the mean blood-oxygen-level dependent (BOLD) signal time series will be extracted for each individual seed-region. Then, the correlation coefficients between the time series of each seed region will be grouped into functional connectivity maps. The functional connectivity maps will be converted into z-scores for normality and used for the statistical analysis. Whole-brain and region of interest functionally connectivity analysis will be conducted.

CONTACTS AND LOCATIONS:
Overall Officials: Andrée-Anne Ledoux, PhD, Principal Investigator — Children's Hospital of Eastern Ontario Research Institute
Locations (1):
- Children's Hospital of Eastern Ontario, Ottawa, Canada

IPD SHARING:
Plan to Share IPD: Yes
We plan to share the study protocol and statistical analysis plan.
Supporting Information: Study Protocol, SAP
Time Frame: These documents will be shared once the protocol is published, approximately 6 months from now.
Access Criteria: The protocol will be accessible online and through Trials.gov.

REFERENCES:
- [Derived] Ledoux AA, Zemek R, Cairncross M, Silverberg N, Sicard V, Barrowman N, Goldfield G, Gray C, Harris AD, Jaworska N, Reed N, Saab BJ, Smith A, Walker L. Smartphone App-Delivered Mindfulness-Based Intervention for Mild Traumatic Brain Injury in Adolescents: Protocol for a Feasibility Randomized Controlled Trial. JMIR Res Protoc. 2024 Apr 11;13:e57226. doi: 10.2196/57226. PMID 38602770